CLINICAL TRIAL: NCT00841464
Title: Prospective Study on the Effect of External Magnetic Stimulation on Patients With Parkinson's Disease
Brief Title: Study on the Effect of External Magnetic Stimulation on Patients With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Parkinson's Disease Research, Education, and Clinical Center, Philadelphia (U.S. Federal Agency)
Collaborators: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 1EA-0000071
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to test the usefulness of external magnetic stimulation (EMS) for treating the motor, cognitive, and neuropsychiatric symptoms of Parkinson's disease (PD).

Participants with Parkinson's disease will be recruited at the PADRECC of the Philadelphia VA Medical Center. Enrolled participants will be randomly assigned to receive either active external magnetic stimulation or fake stimulation. The external magnetic stimulation is delivered by wearing a helmet that is embedded with many small circuits which produce a very small magnetic field around the head. The helmet is to be worn daily for two minutes immediately before bedtime for three months in a row. The helmet is for investigational use only and has not been approved for use by the FDA.

DETAILED DESCRIPTION:
Current research seeks to provide a drug-free, non-invasive and non-toxic therapy for Parkinson's disease through transcranial magnetic stimulation (TMS) in the form of picoTesla magnetic therapy (pTMT). This therapy consists of an electronic device that emits magnetic flux densities that are more than ten million times lower than the magnetic flux density of the earth's magnetic field. Repetitive transcranial magnetic stimulation (rTMS) therapy aims to manipulate overall quality of life by improving motor function, as well as cognitive and neuropsychiatric symptoms such as depression.

ELIGIBILITY:
Inclusion Criteria:

* 40 to 80 years of age
* Diagnosis of possible or probable PD by the UK Brain Bank clinical diagnostic criteria
* Stable anti-Parkinsonian medical regimen for at least 30 days prior to enrollment
* Hoehn & Yahr Scale score of I to III
* No evidence of secondary or atypical Parkinsonism on MRI test in the past year
* Subjects are capable of giving informed consent

Exclusion Criteria:

* Contraindications to MRI (e.g. cardiac pacemaker, claustrophobia, metal fragments or hardware within the orbit or cranium)
* History of stroke or TIA within the past year
* Dementia defined as a MMSE score < 25
* Status post deep brain stimulation surgery
* Unstable medical conditions that would likely prevent the subject from completing the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with Parkinson's disease will be recruited ONLY at the Parkinson's Disease Research, Education, and Clinical Center (PADRECC) of the Philadelphia VA Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-03; Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John E Duda, M.D., Principal Investigator — Parkinson's Disease Research, Education, and Clinical Center (PADRECC), Philadelphia; Timothy Roberts, Ph.D., Principal Investigator — Department of Radiology, The Children's Hospital of Philadelphia
Locations (1):
- Philadelphia VA Medical Center, Philadelphia, Pennsylvania, United States